CLINICAL TRIAL: NCT07026201
Title: Primary Anastomosis After Left Colectomy in Emergency Cases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IBR 00006373
Record Dates: First submitted 2025-04-26; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Complete Obstruction
Keywords: left colon mass
MeSH Terms: conditions — Bites and Stings | interventions — Colectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient with obstructing left colon mass (Other): formal exploration with resection and primary anastomosis
  Interventions: Other: colectomy with primary anastomosis

INTERVENTIONS:
Other: colectomy with primary anastomosis — left hemicolectomy or sigmoidectomy, formal resection was carried out following conventional steps of radical resection.with primary anastomosis
  Other Names: surgical management

SUMMARY:
The aim of this study is to know the outcome of primary anastomosis after left colectomy in emergency cases regarding early post operative complication like surgical site infection , ileus, incidence of leakage, restoration of bowel movement and hospital stay and rate of readmission within one month from the time of intervention.

DETAILED DESCRIPTION:
SPIRIT 2013 Checklist: Recommended items to address in a clinical trial protocol and related documents*

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting to the emergency department with obstructed left colon
* Patients aged between 18 and 80 years old
* Decision of laparotomy is made
* Intraoperative conditions are favorable for anastomosis (e.g., good vascularity, no severe sepsis, no marked tissue edema, no thickened peritoneum)
* Patient agrees to participate in the study

Exclusion Criteria:

* Severe diffuse peritonitis (e.g., peritoneal thickening, thickened bowel loop, severe tissue edema, and pyogenic membrane)
* Marked decreased tissue vascularity due to distension
* Irresectable mass
* Rectal mass
* Patients refusing to participate in the study

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2024-03-20 (Actual); Primary Completion 2024-03-20 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
Incidence of Anastomotic Leakage Within 30 Days Post-Operatively | 30 days after surgery
  * Description: Percentage of patients who develop an anastomotic leak as diagnosed clinically or radiologically
  * Unit of Measure: % of patients
  * Assessment Method: Clinical signs and imaging (e.g., contrast-enhanced CT scan)
Incidence of Surgical Site Infection | 30 days after surgery
  * Description: Percentage of patients who develop a surgical site infection within 30 days after the operation
  * Unit of Measure: % of patients
  * Assessment Method: Clinical evaluation and/or positive wound culture

SECONDARY OUTCOMES:
Incidence of Postoperative Ileus | From date of surgery until first bowel movement, assessed up to 7 days post-surgery
  * Description: Percentage of patients who experience postoperative ileus, defined as absence of bowel movement and need for nasogastric tube beyond 3 days post-surgery
  * Unit of Measure: % of patients
  * Assessment Method: Clinical observation and medical records
Time to Restoration of Bowel Movement | Assessed up to 7 days post-surgery
  * Description: Number of days until first recorded bowel movement after surgery
  * Unit of Measure: Days
  * Assessment Method: Patient report and nursing documentation
Length of Hospital Stay | Assessed up to 14 days post-surgery
  * Description: Total number of days the patient remained in hospital after surgery
  * Unit of Measure: Days
  * Assessment Method: Hospital records
Readmission Rate Within 30 Days | Time Frame: 30 days post-surgery
  * Description: Percentage of patients readmitted to any hospital within 30 days after initial discharge
  * Unit of Measure: % of patients
  * Assessment Method: Patient follow-up and hospital readmission records

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Magid, prof, Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-02-12): https://cdn.clinicaltrials.gov/large-docs/01/NCT07026201/Prot_SAP_ICF_000.pdf